CLINICAL TRIAL: NCT00198471
Title: An Open-label Assessment of Intravitreous Injections of Vitrase (Hyaluronidase for Injection) for Inducing Posterior Vitreous Detachment in Subjects With Moderate to Severe Non-proliferative Diabetic Retinopathy
Brief Title: Assessment of Intravitreous Injections of Vitrase for Inducing Posterior Vitreous Detachment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ISTA-VIT-CS07
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2013-03-15 (Estimated); Status verified 2013-03

CONDITIONS: Vitreous Detachment; Diabetic Retinopathy
MeSH Terms: conditions — Vitreous Detachment; Diabetic Retinopathy | interventions — Chondroitinases and Chondroitin Lyases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vitrase (Experimental): A single intravitreous injection of Vitrase 93 USP Units (75 IU) on Study Day 1.
  Interventions: Drug: Vitrase

INTERVENTIONS:
Drug: Vitrase
  Other Names: ovine hyaluronidase

SUMMARY:
The purpose of this study is to assess the efficacy of intravitreous injections of Vitrase to induce posterior vitreous detachment(PVD) in subjects with moderate to severe non-proliferative diabetic retinopathy.

ELIGIBILITY:
Inclusion Criteria:

* Moderately severe to severe non-proliferative diabetic retinopathy
* Best Corrected Visual Acuity (BCVA) in Early Treatment Diabetic Retinopathy Study (ETDRS) with pinhole of 20/320 or better in study eye & 20/50 or better in non-study eye.

Exclusion Criteria:

* Contraindications or hypersensitivities to Vitrase or anesthesia
* Any significant illness that could be expected to interfere with trial
* Prior Vitrase therapy
* Either a past diagnosis of clinically significant macular edema (CME) in study eye that required treatment or current CME that may require focal laser treatment within the next 30 days
* For either eye: ongoing ocular infection, inflammation or history of herpetic corneal lesion; an intravitreous injection within 30 days; glaucoma; intraocular pressure (IOP) of less than 5mmHg; retinal detachment or ocular tumors
* For study eye: vascular occlusive disease of fundus; corneal, lenticular or ocular media abnormalities; a significant ocular trauma within 6 months; previous vitrectomy; any prior laser treatment, cryo-retinopexy or any intraocular surgery; either a partial or complete posterior vitreous detachment (PVD); myopia of 6 or more spherical diopters and/or axial length exceeding 26mm; significant retinal pathology

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10
Dates: Start 2005-07; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Vitreous detachment | Day 28
  The proportion of subjects achieving a complete posterior vitreous detachment by Study Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Jon Williams, PhD, Study Director — ISTA Pharmaceuticals, Inc.
Locations (4):
- United States (4):
  - Edgar L. Thomas, MD, Beverly Hills, California
  - Ronni Lieberman, MD, New York, New York
  - Valley Retina Institute, PA, McAllen, Texas
  - The Virginia Retina Center, Leesburg, Virginia